CLINICAL TRIAL: NCT06200337
Title: The Change in Cutaneous Temperature When Using Acupuncture at Zhongzhu (TB-3) and Shugu (BL-65) Acupoints in Healthy Participants: A Pilot, Randomized, Double-blind, Self-controlled Trial
Brief Title: The Change in Cutaneous Temperature When Using Acupuncture at TB-3 and BL-65 Acupoints in Healthy Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loc Cong Dai Tran, MD (Other)
Collaborators: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Sponsor-Investigator, Loc Cong Dai Tran, MD, Principal Investigator, School of Medicine - Vietnam National University at Ho Chi Minh city
Organization: School of Medicine - Vietnam National University at Ho Chi Minh city (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 1064/HĐĐĐ-ĐHYD
Record Dates: First submitted 2023-12-05; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-12

CONDITIONS: Healthy Participants
Keywords: acupuncture; skin surface temperature

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants: They did not know about acupuncture, meridian theory, and acupoints. The investigator informs the information about the specific location of the acupoints used and the purpose of the study. The investigator provided a questionnaire to assess the participants' knowledge of meridian and acupressure theory, expectations, and motivation to participate.
  Infrared image analyst: The person analyzing the infrared images is not familiar with acupuncture methods. We trained them for two weeks on using FLIR Thermal Studio software and identifying experimental skin areas. After analysis, the infrared image analyst encodes the data and sends it back to the data analyst.
  Data analyst: The investigator analyzed the data and was not involved in the randomization and data collection stages.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Other): In the first session, acupuncture was applied at BL65, the second at TB3, and the third at SP3. Each session was seperated 24 hours interval.
  Interventions: Procedure: Fine needle acupuncture
- Group B (Other): In the first session, acupuncture will be applied at SP3, the second at BL65, and the third at TB3. Each session was seperated 24 hours interval.
  Interventions: Procedure: Fine needle acupuncture
- Group C (Other): In the first session, acupuncture will be applied at TB3, the second at SP3, and the third at BL65. Each session was seperated 24 hours interval.
  Interventions: Procedure: Fine needle acupuncture

INTERVENTIONS:
Procedure: Fine needle acupuncture — All participants underwent three 24-hour apart sessions. In each session, the acupuncturist inserted two sterile needles into the left and right acupoints with a 90-degree angle and 0.5 to 1 cun in depth for TB3, 0.3 to 0.5 cun for BL65, and 0.3 to 0.5 cun for SP3. The acupuncturist rotated the needle at an angle of 180-270 degrees within 1 minute, with a frequency of 60 - 120 times/minute for stimulation.

SUMMARY:
For more than 2,500 years, traditional medicine, especially acupuncture, has been widely used in health care and recognized by the World Health Organization (WHO) to manage various diseases. Besides, many molecular biological mechanisms of acupuncture in pain management have been elucidated. Acupuncture is a safe, effective, and cost-effective therapy, reducing the overuse of opioid pain relievers. In neck pain treatment, many clinical studies used remote acupoints, which have specific effects on the neck. Among them, the Stream points in the Five Stream acupoints system are the most used acupuncture points in the treatment of neck pain. However, the relationship between these acupoints and the neck has not been proven. The goal of this trial is to compare the change in skin surface temperature at the neck and the cutaneous zone before and after using acupuncture at the control acupoint (SP3) and two research acupoints (TB3 and BL65) in healthy volunteers. The main questions it aims to answer are:

* Whether the Zhongzhu and Shugu acupoints change the skin temperature in the neck area?
* How does the change in temperature correlate with the cutaneous zone distribution of the Shaoyang and Taiyang meridians, respectively?

DETAILED DESCRIPTION:
Participants and Methods: The change in skin surface temperature before and after acupuncture at the control acupoint (SP3) and two research acupoints (TB3 and BL65) in healthy volunteers will be compared in a randomized, double-blinded, self-controlled trial. A total of 30 participants will be assigned to 3 groups (A, B, and C), and the allocation will be 1:1:1. Every group will go through three trial stages spaced out by 24 hours, with each stage corresponding to one acupoint on both sides. Group A: In the first trial stage, acupuncture will apply at BL65, the second trial stage at TB3, and the third trial stage at SP3. Group B: In the first trial stage, acupuncture will apply at SP3, the second stage at BL65, and the third stage at TB3. Group C: In the first trial stage, acupuncture will apply to participants at TB3, the second stage at SP3, and the third stage at BL65. The primary outcome of acupuncture at the TB3, BL65, and SP3 acupoints will be the alteration in skin surface temperature at the neck area and the cutaneous zone. The skin surface temperature was measured by an Infrared Thermal Camera brand FLIR C5 and thermal images were analyzed by FLIR Thermal Studio software.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants.
* BMI: 18.5 - 23 kg/m2
* Mental alertness, good contact, cooperation with researchers.
* Having no psychiatric stress problem during acupuncture day (confirmed by answering the DASS21 questionnaire with stress points less than 15 points).
* Vital signs within normal limits:

  * Heart rate from 60 to 99 beats per minute.
  * Systolic blood pressure between 90 and 139 mmHg.
  * Diastolic blood pressure between 60 and 89 mmHg.
  * Body temperature: 36.59 ± 0.43 degrees Celsius.
  * Breathing rate: 16 ± 3 breaths per minute.
* Having no disease or using drugs which may change the body temperature.
* Not currently participating in other intervention studies.
* Volunteers who agree to participate and sign the Informed Consent Form, following a detailed explanation of clinical trials.
* Having no acupuncture knowledge yet.

Exclusion Criteria:

* Participate in vigorous physical activities 2 hours before the procedure.
* Taking stimulants (alcohol, beer, coffee, and tobacco) within 24 hours before participating the study.
* Staying up late at night or having a sleep disorder before the procedure
* Women who were in menstruation period, pregnancy, or breastfeeding.
* Having skin injuries, dermatitis-skin infections, or wounds in the area to be investigated.
* Applying chemical or pharmaceutical products to the site of the skin to be investigated before participating the study.
* Using physical therapy, heat therapy, cupping therapy, massage, and acupuncture on the site of the skin to be investigated within 24 hours before participating the study.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
The change in skin surface temperature at the neck | Five time points: baseline; 6 minutes (after needled and fisrt rotation); 12 minutes (after second rotation); 17 minutes (after rejection); and 22 minute
  The change in skin surface temperature (in degree Celsius) at the neck area when using acupuncture at Zhongzhu (TB3) and Shugu (BL65), in comparison with Taibai (SP3).
The change in skin surface temperature at the cutaneous zone of Taiyang and Shaoyang meridians | Five time points: baseline; 6 minutes (after needled and fisrt rotation); 12 minutes (after second rotation); 17 minutes (after rejection); and 22 minute
  The change in skin surface temperature (in degree Celsius) at the cutaneous zone of the Taiyang meridian compared with the Shaoyang meridian when using acupuncture at Zhongzhu (TB3) and Shugu (BL65).

SECONDARY OUTCOMES:
Adverse effects | During and 7-day after procedure
  Investigating the adverse events (in percentage) when using acupuncture at Zhongzhu (TB3), Shugu (BL65), and Taibai (SP3) acupoints
The adaptation to acupoints effects | Five time points: baseline; 6 minutes (after needled and fisrt rotation); 12 minutes (after second rotation); 17 minutes (after rejection); and 22 minute
  Comparision of the change in skin surface temperature (in degree Celsius) at the neck between 3 groups when using acupuncture at Zhongzhu (TB3), Shugu (BL65), Taibai (SP3), respectively

OTHER OUTCOMES:
Blood pressure | Baseline and 5 minutes after needle rejection
  Comparison of the blood pressure in mmHg when acupuncture at Zhongzhu (TB3), Shugu (BL65), Taibai (SP3).
  Comparison of the blood pressure, heart rate, body temperature, and skin surface temperature at the neck before acupuncture at Zhongzhu (TB3), Shugu (BL65), Taibai (SP3).
Pulse rate | Baseline and 5 minutes after needle rejection
  Comparison of the pulse rate in rate per minute when acupuncture at Zhongzhu (TB3), Shugu (BL65), Taibai (SP3).
Body temperature | Baseline and 5 minutes after needle rejection
  Comparison of the body temperature in degree Celsius when acupuncture at Zhongzhu (TB3), Shugu (BL65), Taibai (SP3).

CONTACTS AND LOCATIONS:
Overall Officials: Bay Thi Nguyen, MD., PhD., Study Director — University of Medicine and Pharmacy at Ho Chi Minh City
Locations (1):
- School of Medicine, Vietnam National University at Ho Chi Minh City, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Demographic characteristic and outcome data will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 3 months and ending 1 years after the publication of results

REFERENCES:
- [Background] Molsberger AF, Manickavasagan J, Abholz HH, Maixner WB, Endres HG. Acupuncture points are large fields: the fuzziness of acupuncture point localization by doctors in practice. Eur J Pain. 2012 Oct;16(9):1264-70. doi: 10.1002/j.1532-2149.2012.00145.x. Epub 2012 Apr 10. PMID 22492604
- [Background] Huang T, Huang X, Zhang W, Jia S, Cheng X, Litscher G. The influence of different acupuncture manipulations on the skin temperature of an acupoint. Evid Based Complement Alternat Med. 2013;2013:905852. doi: 10.1155/2013/905852. Epub 2013 Feb 13. PMID 23476709
- [Background] Ots T, Kandirian A, Szilagyi I, DiGiacomo SM, Sandner-Kiesling A. The selection of dermatomes for sham (placebo) acupuncture points is relevant for the outcome of acupuncture studies: a systematic review of sham (placebo)-controlled randomized acupuncture trials. Acupunct Med. 2020 Aug;38(4):211-226. doi: 10.1177/0964528419889636. Epub 2020 Feb 6. PMID 32026725
- [Background] Amalu W, Block J, Chaudhry A. International academy of clinical thermology quality assurance guidelines. Standards and protocols in clinical thermographic imaging. Current Revision July 2015; July 2018. 2021.
- [Background] Guan L, Li G, Yang Y, Deng X, Cai P. Infrared thermography and meridian-effect evidence and explanation in Bell's palsy patients treated by moxibustion at the Hegu (LI4) acupoint: Overall regulation or a specific target? Neural Regen Res. 2012 Mar 25;7(9):680-5. doi: 10.3969/j.issn.1673-5374.2012.09.007. PMID 25745463
- [Background] Mo MJ, Hwang DR, Lee JH, et al. Analysis on the Acupuncture Contents of the Domestic Neck Pain and HIVD-Cervical Spine Clinical Studies: a literature review. 2017;34(2):113-125.